CLINICAL TRIAL: NCT04083469
Title: Identifying Student Opinion Leaders to Lead E-cigarette Interventions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 resulted in school closures.
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Kar-Hai Chu, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY19040095
Record Dates: First submitted 2019-08-19; First posted 2019-09-10 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: E-Cig Use; Adolescent Behavior
MeSH Terms: conditions — Vaping; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Investigators will conduct a social network survey for 6th graders. Students will be asked to identify their close peers based on several dynamics: friendship, opinion leadership, academic support, and personal support. Social network analyses will identify opinion leaders based on network centrality measures. Surveys will be administered before and after the intervention.
  Investigators will adapt modules from CATCH My Breath, an evidence-based e-cigarette intervention supported by University of Texas and MD Anderson Cancer Center. The 8 schools will be randomized to receive the intervention led by either (1)an adult content-expert or (2)a peer-nominated opinion leader to students who nominated them or (3)a peer-nominated opinion leader to students who did not nominate them. Primary outcomes will be acceptability and feasibility measures, including (1)recruitment and (2)retention rates. Secondary outcomes will include intention-to-use e-cigarettes and knowledge about e-cigarettes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer-Led Peer-Elected Intervention (Experimental): The e-cigarette intervention program will be administered to students by an elected peer leader. The audience will consist of students that nominated the peer-leader.
  Interventions: Behavioral: Peer-Led Peer-Elected Intervention
- Adult-Led Intervention (Other): The e-cigarette intervention program will be administered to students by an adult educator.
  Interventions: Behavioral: Adult-Led Intervention
- Peer-Led Non-Elected Intervention (Other): The e-cigarette intervention program will be administered to students by an elected peer leader. The audience will consist of students that nominated a different peer-leader.
  Interventions: Behavioral: Peer-Led Non-Elected Intervention

INTERVENTIONS:
Behavioral: Peer-Led Peer-Elected Intervention — The intervention will be given to students by a peer opinion leader that the students in the audience elected. The intervention is a version of CATCH My Breath curriculum that has been modified to facilitate peer leadership.
  Arms: Peer-Led Peer-Elected Intervention
Behavioral: Adult-Led Intervention — The intervention will be given to students by an adult. The intervention is a version of CATCH My Breath curriculum that has been modified to match the Peer-Led Intervention curriculum but is able to be administered by an adult.
  Arms: Adult-Led Intervention
Behavioral: Peer-Led Non-Elected Intervention — The intervention will be given to students by a peer opinion leader that was elected by other students. The intervention is a version of CATCH My Breath curriculum that has been modified to facilitate peer leadership.
  Arms: Peer-Led Non-Elected Intervention

SUMMARY:
This research will explore the feasibility of leveraging social network analysis to identify 6th grade opinion leaders to lead a school-based e-cigarette intervention. The project will be conducted for 6th graders in 8 schools in the Pittsburgh area.

DETAILED DESCRIPTION:
Specific Aim 1: Participants will be recruited from 8 Pittsburgh-area schools. The investigators will conduct a social network survey for all 6th graders in each school. Students will be asked to identify their closest peers based on several relationship dynamics: friendship, opinion leadership, academic support, and personal support.

Specific Aim 2: The investigators will adapt modules from CATCH My Breath, an evidence-based, school-implemented e-cigarette intervention supported by University of Texas and MD Anderson Cancer Center. The 8 schools will be randomized to receive the intervention led by either (1) an adult content-expert or (2) a peer-nominated opinion leader to students who nominated them or (3) a peer-nominated opinion leader to students who did not nominate them. Surveys will be administered before and after the intervention. Primary outcomes will be acceptability and feasibility measures, including (1) recruitment and (2) retention rates. Secondary outcomes will include e-cigarette use, intention-to-use e-cigarettes, and knowledge about e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* 6th grade student at Linton, Founder's Hall, Woodland Hills, Steel Valley, Greensburgh Salem, Freedom, Marion, or Rostraver schools

Exclusion Criteria:

* Students who are unable to read the surveys will be excluded from data collection. However, all students will still participate in the e-cigarette program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability: follow-up survey | 5 months
  Acceptability of the intervention will be assessed via the follow-up survey administrated to students following the program.
  1. Do you feel the lessons were appropriate for the subject?
  2. Were you confident in the person conducting the lesson?
  Questions will be measured in a 5 point Likert scale.
Feasibility: recruitment and retention rates | 5 months
  Feasibility of the intervention will be assessed via the recruitment and retention rates.
  1. Recruitment = number of students who agree to participate / number of students in school
  2. Retention = number of students who completed the program / number of students who began the program

SECONDARY OUTCOMES:
Intention-to-use and knowledge about e-cigarettes (based on National Youth Tobacco Survey) | 5 months
  Intention-to-use and knowledge about e-cigarettes will be assessed via the e-cigarette survey that will be administered after the program. Measures are adapted from the National Youth Tobacco Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Kar-Hai Chu, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Chu KH, Matheny S, Furek A, Sidani J, Radio S, Miller E, Valente T, Robertson L. Identifying student opinion leaders to lead e-cigarette interventions: protocol for a randomized controlled pragmatic trial. Trials. 2021 Jan 6;22(1):31. doi: 10.1186/s13063-020-04990-z. PMID 33407805